CLINICAL TRIAL: NCT00753493
Title: Phase I Pharmacokinetic and Safety Study of Intravenous Topiramate in Adult Patients
Brief Title: Pharmacokinetics and Safety of Intravenous Topiramate in Adult Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0804M29861
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Epilepsy; Migraines
MeSH Terms: conditions — Epilepsy; Migraine Disorders | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): This is a one arm pharmacokinetic and safety study.
  Interventions: Drug: intravenous topiramate

INTERVENTIONS:
Drug: intravenous topiramate — Single 25 mg IV dose given in addition to subject's normal morning dose of topiramate
  Other Names: Topamax

SUMMARY:
The aims of this study are to determine, in adult patients on maintenance topiramate therapy, the steady-state pharmacokinetics and safety of orally and intravenously administered topiramate.

DETAILED DESCRIPTION:
The long-term goal of this research project is to develop a more effective, safer therapy for neonatal seizures. Prior to using an investigational intravenous topiramate formulation in children and neonates, the pharmacokinetics and safety of the formulation must be demonstrated in adults. The immediate aims of this study are to determine the pharmacokinetics and safety of a novel intravenous topiramate formulation. An additional aim is to determine if sex, advancing age, or genotype affects topiramate absorption, distribution, or elimination.

ELIGIBILITY:
Inclusion Criteria:

* Persons taking topiramate
* Persons 18 years of age and older

Exclusion Criteria:

* Patients who are pregnant
* Patients who are breast feeding
* Patients with significant medical problems who may not tolerate intravenous administration
* Patients taking medications known to affect topiramate disposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Safety as measured by the occurrence of adverse events | 96 hours after dosing
  Occurrence of adverse events in the 4 days following Topiramate dose

CONTACTS AND LOCATIONS:
Overall Officials: James C Cloyd, PharmD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States